CLINICAL TRIAL: NCT00886990
Title: Comparing the Efficacy and Safety of Single Versus Double Ritonavir-boosted Protease Inhibitor (PI)-Based Antiretroviral Therapy (ART) Regimens for Children Failing Non Nucleoside Reverse Transcriptase Inhibitor (NNRTI)-Based Treatment
Brief Title: Efficacy and Safety of Single Versus Double Ritonavir-boosted Protease Inhibitor (PI)-Based Antiretroviral Therapy (ART) Regimens
Status: Completed | Type: Observational
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: Ministry of Education, Thailand (Other)
Responsible Party: Sponsor
Other Study IDs: HIV-NAT 086
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: HIV Infection; HIV Infections
Keywords: single- and double-boosted PI; second line regimen; NNRTI failure; HIV-infected children; Compare virological efficacy and safety of single- or double-boosted PI regimens as second line therapy in children with NNRTI-based treatment failure; treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — Ritonavir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Receiving a single PI boosted by low dose ritonavir
  Interventions: Drug: ritonavir-boosted PI-based second line treatments
- 2: Receiving two PIs boosted by low dose ritonavir or one PI plus full dose ritonavir
  Interventions: Drug: two PIs boosted by low dose ritonavir or one PI plus full dose ritonavir

INTERVENTIONS:
Drug: ritonavir-boosted PI-based second line treatments — single PI boosted by low dose ritonavir
  Groups: 1
Drug: two PIs boosted by low dose ritonavir or one PI plus full dose ritonavir — two PIs boosted by low dose ritonavir or one PI plus full dose ritonavir
  Groups: 2

SUMMARY:
The virological efficacy will be no different in children treated with single versus double boosted PI second line ART regimens.

DETAILED DESCRIPTION:
A total of 50,620 Thai children have been diagnosed with HIV infection in Thailand between 1988 and 2005, of whom only 20,000 are still living.1 The production of generic ART by the Thai Government Pharmaceutical Organization (GPO), which began in 2002 has given the Thai Government the ability to offer highly active antiretroviral therapy for all children.2 As of June 2006, there were over 6000 children receiving ART within the government program, and it is estimated that another 1500 children are receiving care in the private sector.1

The Thai National Access to Care program provides two nucleoside reverse transcriptase inhibitors (NRTIs) and one NNRTI as the first-line regimen of choice. The most commonly used regimen is GPO-vir S, which has been shown to have acceptable pharmacokinetic parameters3 and excellent treatment outcome4. A study of 107 children on NNRTI-based treatment, including half with GPO-vir S, showed that despite their low baseline CD4 of 3% and high viral load of 5.4 log, the children had excellent virological response, with 76% having HIV RNA below 50 copies/ml at week 72.4 In another study of 192 children with advanced HIV disease, the hospitalization rate decreased from 31% during the first six months to 2% at three years after HAART. The mortality rate decreased from 6% during the first six months of HAART to less than 1% after that.5

Nevertheless, Thailand is faced with growing numbers of children experiencing failure on NNRTI-based regimens as 20% or more are expected to fail based on published literature4, 6. This could result in 1000 or more Thai children needing to change therapy in the new future. Therefore, there is an urgent need to find appropriate second line treatments.

Developed and developing countries guidelines recommend regimens with a single PI plus low-dose ritonavir boosting (boosted PI) in combination with 2 NRTIs for adults and children failing NNRTI-based treatments.6-8 There is limited data on the antiviral efficacy of boosted PI second line treatment following failure from PI-sparing first line regimens. As the success of second line PI regimens in PI-experienced patients depends heavily on the number of PI mutations present9, 10, it is reasonable to assume that in NNRTI failures without any PI mutations, most of the patients will do well. However, this also depends on the number of active NRTIs that can be used in the second line regimens. Meta-analysis has shown that NNRTI failures tend to be associated with more NRTI mutations than PI failures.11 This is particularly true in developing countries where switching to second line therapy usually occur when there is late virological failure, and patients show signs of clinical and/or CD4 failure.12 A high likelihood of multi-NRTI resistance coupled with limited NRTIs choices can render the second line regimens less active. In these circumstances, it is unclear how effective a single boosted PI with recycle NRTIs second line treatment would be. Therefore, double boosted PIs with or without NRTIs have been proposed as a second line option in the 2007 Ministry of Public Health Treatment Guidelines for children with HIV infection.13 The pharmacokinetic enhancement of 2 different PIs with low-dose ritonavir offers a unique benefit in maintaining a high genetic barrier to resistance.

There are few choices for second-line therapy in children. Lopinavir/ritonavir is the PI of choice because it is the only ritonavir-co-formulated drug and the only liquid PI. It also has excellent efficacy in trials of single-boosted PI in children.14, 15 Indinavir is a commonly used PI in Thailand as it is the least expensive PI. Plipat N, et al. showed evidence supporting the efficacy, safety and pharmacokinetics of a lower dose of 230-300 mg/m2 indinavir boosted with ritonavir and used in combination with 2NRTIs in Thai children.16 The efficacy of double boosted PI, saquinavir/lopinavir/ritonavir, was investigated in 50 children with NRTI/NNRTI failure. The regimen was effective: 80% and 60% had HIV RNA below 400 and 50 copies/ml respectively at week 48. However, the regimen was burdensome because of the large pill sizes, and the occurrence of hyperlipidaemia in 44% of children at week 48 caused concern 17, 18 Fortunately, no failing children were found to have PI mutations.19 A small study in Caucasian adults using the same regimen also show good efficacy.20

ELIGIBILITY:
Inclusion Criteria:

1. Children (< 18 years old) with HIV infection
2. Have failed NNRTI-based ART
3. Received second-line regimen with either one or two boosted PIs (Note: low dose ritonavir to boost the other PI will not be count as additional PI)
4. Began ritonavir-boosted PI prior to June 30, 2007

Exclusion Criteria:

1. Have previously received PI treatment for longer than 30 days prior to the current PI regimen.
2. Has previously or currently been treated with abacavir or tenofovir
3. Currently on ART other than NRTI, NNRTI and PI drug classes

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Data of children who satisfy the following eligibility criteria will be included.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2007-10; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Primary endpoint will be the proportions of subjects with HIV RNA below 400 and 50 copies/ml over a 48-week period. | 48 weeks

SECONDARY OUTCOMES:
HIV/AIDS disease progression, changes in CD4+ cell count or percentage, treatment failure, antiretroviral drug resistance, serious adverse events, grade 3 or grade 4 events, and toxicities | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thanyawee Puthanakit, MD, Principal Investigator — The HIV Netherlands Australia Thailand Research Collaboration; Jintanat Ananworanich, MD, Ph.D, Principal Investigator — The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) and South East Asia Research Collaboration with Hawaii (SEARCH), The Thai Red Cross AIDS Research Centre, Bangkok
Locations (8):
- Thailand (8):
  - Petchburi Hospital, Petchburi, Petchburi
  - HIV-NAT, Bangkok
  - Queen Sirikit National Institute of Child Health, Bangkok
  - Siriraj Hospital, Mahidol University, Bangkok
  - Department of Pediatrics, Faculty of Medicine, Chiang Mai University Hospital, Chiang Mai
  - Chiang Rai Regional Hospital, Chiang Rai
  - Khon Kaen University, Khon Kaen
  - Bamrasnaradura Institute, Nonthaburi

REFERENCES:
- See also: HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org